CLINICAL TRIAL: NCT06199024
Title: The Effect of Cinnamon Supplementation on Infertility Treatment Outcomes in Infertile Women With Polycystic Ovary Syndrome (PCOS) Candidate of in Vitro-fertilization (IVF): A Pilot Double Blind Randomized Controlled Clinical Trial
Brief Title: Cinnamon and COH in PCOS Women Underdoing IVF/ICSI Cycles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 402000037; IRCT20080831001141N44 (Other: https://www.irct.ir/)
Record Dates: First submitted 2023-11-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon supplementation (Experimental): In intervention group patients will take 1500 mg daily (3 tablets of cinnamon 500 mg, Sagepad Darou Pharmaceutical Company, Iran) that is, 4 weeks before the start of the new IVF cycle and 2 weeks during the ovarian stimulation process.
  Interventions: Dietary Supplement: Oral cinnamon supplementation
- Control group (Placebo Comparator): Patients take 3 placebo pills daily (containing white wheat flour, which is similar to cinnamon pills in terms of size, shape, color and smell, Sagepad Darou Pharmaceutical Company, Iran) 4 weeks before starting the ovarian stimulation/in vitro fertilization (COS/IVF) cycle and 2 weeks during the ovarian stimulation procedure, the ovary will be stimulated
  Interventions: Dietary Supplement: Oral cinnamon supplementation

INTERVENTIONS:
Dietary Supplement: Oral cinnamon supplementation — In intervention group patients will take 1500 mg daily (3 tablets of cinnamon 500 mg, Sagepad Darou Pharmaceutical Company, Iran) that is, 4 weeks before the start of the new IVF cycle and 2 weeks during the ovarian stimulation process.

SUMMARY:
In patients with polycystic ovary syndrome, insulin resistance increases, and since the extracts from cinnamon reduces insulin resistance by two mechanisms (1- increasing activation of the IRS/PI-3 kinase insulin signaling pathway and 2- stimulate auto phosphorylation of the insulin receptor and inhibit protein tyrosine phosphatase I). Through these two mechanisms cinnamon extract make adipocytes to increase the glucose uptake and glycogen synthesis. So this hypothesis arises that it can be effective in improving the symptoms of polycystic ovary syndrome.

DETAILED DESCRIPTION:
This double-blind randomized clinical trial will be conducted in Royan Institute on patients with polycystic ovary syndrome undergoing in vitro fertilization cycle treatment to evaluate the effect of Cinnamon supplementation during controlled ovarian stimulation in patients with polycystic ovary syndrome.PCOS cases were diagnosed based on the Rotterdam criteria (4), and the presence of at least two of the following criteria: menstrual irregularity (cycle length <26 days or >35 days or variation between consecutive cycles of >10 days); clinical (presence of hirsutism evaluated by a Ferriman- Gallwey score >8, severe acne and alopecia) or biochemical (total testosterone concentration >0.5 ng/ml and/or free testosterone>3.5 pg/ml) hyperandrogenism; or ultrasound evidence of polycystic ovaries. Hirsutism was assessed according to the Ferriman-Gallwey-score and examination of nine body areas for coarse terminal hair, including upper lip, chin and chest, upper and lower areas of the abdomen, thighs and upper arms. In each part, the severity of hirsutism was graded from 1 to 4 and the participants with the total score of 8 and above considered as having hirsutism. PCOM was defined as the presence of 12 or more ovarian cysts with 2-10 mm diameter per ovary and/or ovarian volume ≥10 cm3. Vaginal ultrasound was performed by an ultrasound specialist and radiologist using an Aloka α-10 with a transvaginal 6-7.5 MHz probe (Medison Co., Japan).

The controlled ovarian stimulation method will be the same in all participants using the standard antagonist protocol. All patients diagnosed with polycystic ovary syndrome who are eligible based on the Rotterdam criteria and other inclusion and exclusion criteria stated in the general information section of the clinical trial and who have written consent to participate in the study will be examined. Patients will be randomly assigned into two groups using the block method in a size of 6, and each person will be given an exclusive code to keep the allocation hidden. The details of random allocation in terms of drug and placebo grouping are solely at the disposal of the project's pharmacist colleague, who have no role in the process of sampling and follow-up of patients.The medicine packages, as well as the appearance and smell of cinnamon and placebo tablets, are completely similar to each other. The methodologist prepared the drugs based on the block randomization method and prepared the coded list and put an English three-letter code label on the medicine cans. When an eligible patient is referred to a clinical physician, the principal investigator provides him with an envelope containing a drug code based on a randomized list, and the drug package with the same code is delivered to the patient. In this way, the patient and the clinical doctor following the patient will not know the type of drug (cinnamon or placebo).The method of ovarian stimulation and placebo consumption in the control group will be completely similar to the intervention group. In the intervention group, women will take 1500 mg daily (3500 mg cinnamon tablets, Sagepad Darou Pharmaceutical Company, Iran) that is, 4 weeks before the start of the new IVF cycle and 2 weeks during the ovarian stimulation process. Control group: patients take 3 placebo pills daily (containing white wheat flour, which is similar to cinnamon pills in terms of size, shape, color and smell, Sagepad Darou Pharmaceutical Company, Iran) 4 weeks before starting the ovarian stimulation/in vitro fertilization (COS/IVF) cycle and 2 weeks during the ovarian stimulation procedure, the ovary will be stimulated. Total number of retrieved oocytes and total number of MII oocytes will be compared between groups as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with polycystic ovary syndrome (PCOS) diagnosed according to the Rotterdam criteria who meet at least 2 of the following three criteria including: (1) oligomenorrhea or anovulation, (2) hyperandrogenism (clinical or biochemical ng/ dL 80 ≤ serum T level), (3) the presence of polycystic ovaries in ultrasound).
* The age range of 18 to 38 year.
* Written consent to participate in the study

Exclusion Criteria:

* Body mass index above 35 kg/m2
* Chronic and Endocrine disorders including diabetes mellitus, hyperprolactinemia, hypertension, Cushing's syndrome
* Autoimmune disorders
* History of recurrent pregnancy loss
* Genital, ovarian or uterine abnormalities
* Hydrosalpinx diagnosis
* Congenital adrenal hyperplasia, androgen-producing tumors or acromegaly
* Sensitivity to cinnamon
* Daily and frequent consumption of cinnamon to treat infertility
* Severe male factor infertility
* Moderate to severe endometriosis diagnosis Use of other hypoglycemic, insulin-sensitizing drugs (e.g. Metformin) or other antioxidant supplement (e.g. Myo-inositol) and β-blocker before or during the study

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | 32-34 hours after hCG administration (approximately 6 weeks after intervention)
  At the point of ovum pick-up, the total number of retrieved oocytes is counted by the embryologist. Therefore, it will be possible to measure the results one hour after oocytes retrieval.
Total number of mature (MII) oocytes | 32-34 hours after hCG administration (approximately 6 weeks after intervention)
  At the point of ovum pick-up, the total number of retrieved oocytes is counted by the embryologist. Therefore, it will be possible to measure the results one hour after oocytes retrieval.
Oocyte recovery ratio | 32-34 hours after hCG administration (approximately 6 weeks after intervention)
  This ratio is obtained by dividing the total number of retrieved oocytes by the total number of aspirated follicles from both ovaries.
Oocyte maturity rate | 32-34 hours after hCG administration (approximately 6 weeks after intervention)
  This ratio is calculated by dividing the number of mature oocytes (MII) obtained by the total number of retrieved oocytes from both ovaries.

SECONDARY OUTCOMES:
Fertilization rate | 17-18 h after intracytoplasmic sperm injection and/or in-vitro insemination by checking the number of polar bodies and pronuclei
  The fertilization rate is defined as the ratio between the number of diploid zygotes and the number of mature oocytes
Quality of obtained embryos | 3 days after intracytoplasmic sperm injection or in vitro fertilization (IVF/ICSI) procedure
  Embryo grade is assessed under an inverted microscope 3 days after the intracytoplasmic sperm injection procedure. The quality of embryos is graded from 1 to 3 under inverted microscope 3 days after the intracytoplasmic sperm injection procedure. Embryos with even-sized blastomeres and/or ≤10% fragments is classified as Grade 1 (Excellent or good quality). Grade 2 embryos (moderate or fair quality) have blastomeres with slightly-moderate size differences and/or 10- 20% fragments. Grade 3 embryos (poor quality) have markedly different-sized blastomeres and/or >20% fragments.

CONTACTS AND LOCATIONS:
Overall Officials: Parvaneh Afsharian, Ph.D, Study Chair — Royan Institute; Zeynab Siahnouri, Doctor, Study Director — Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran